CLINICAL TRIAL: NCT04050332
Title: Can RFID Technology Capture Stair Walking: A Pilot Study
Brief Title: Can RFID Technology Capture Stair Walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Jennifer Gay, Associate Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROJECT00000674
Record Dates: First submitted 2019-08-02; First posted 2019-08-08 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Physical Activity; Blood Pressure
Keywords: Radio Frequency Identification Device
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stair Walking (Experimental): Participants in this arm will engage in four minutes of stair walking while being tracked by radio frequency identification equipment.
  Interventions: Behavioral: Stair Walking
- Control (No Intervention): Participants in this arm will stand in the stairwell for four minutes while being tracked by radio frequency identification equipment.

INTERVENTIONS:
Behavioral: Stair Walking — Walking up and down stairs for four minutes at a comfortable pace
  Arms: Stair Walking

SUMMARY:
There are two main aims for this study:

1. conduct a proof-of-concept study illustrating how radio-frequency identification technology can be used to document the timestamps and duration of stair walking (ascending and descending stairs), and detect if an individual is stationary in the stairwell.
2. assess the association of a 4-min bout of self-paced stair walking with changes in blood pressure, mood, and perceived exertion.

DETAILED DESCRIPTION:
Objective, passive methods for measuring physical activity participation can minimize error associated with self-report bias and cognitive processing. This study will test the utility of radio frequency identification (RFID) for the measurement of stair walking within buildings. RFID readers will be placed at stairwell entrances on each floor. Participants will wear a RFID tag. As the participant walks past the different readers going up and down the stairs, the reader will log the date and time. The frequency and duration of time in the stairwell can be calculated, as can an estimated speed.

There are known effects for blood pressure (hypotensive) and moodafter exercise. However, few studies have assessed this effect for short bouts (<10 minutes) of exercise. Participants will have their pre- and post-stair walking blood pressure measured to determine the hypotensive and mood enhancing effects of four minutes of stair walking at a comfortable pace. Participants also will rate the exertion level of four minutes of stair walking at a self-selected pace.

ELIGIBILITY:
Inclusion Criteria:

* in desired age range

Exclusion Criteria:

* Unable to or uncomfortable climbing stairs
* Not cleared for exercise using the Physical Activity Readiness Questionnaire (PAR-Q+)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Stair walking duration | Calculated after the completion of the 4-minute stair walking episode
  Duration, in seconds, of stair walking as tracked by the RFID equipment
Stair walking distance | Calculated after the completion of the 4-minute stair walking episode
  Distance, in number of stairs climbed, as tracked by the RFID equipment
Stair walking speed | Calculated after the completion of the 4-minute stair walking episode
  Speed of stair walking, in stairs per second based on duration and distance, as tracked by the RFID equipment

SECONDARY OUTCOMES:
Blood Pressure | Before stair walking and 2-minutes and 5-minutes post stair walking
  Systolic and diastolic blood pressure
Borg's Rating of Perceived Exertion | Immediately after stair walking
  A one-item measure of a participant's perceived physical effort during an activity. Responses range from 6 (no exertion) to 20 (maximal exertion), where higher scores indicate a greater perceived exertion.
Mental Energy | Before and immediately after stair walking
  Measured by self-report using the State Energy and Fatigue Scale. There are 3 items, scored using a number line from 0 to 100, that are summed to generate a score, where higher scores indicate greater mental energy.
Mental Fatigue | Before and immediately after stair walking
  Measured by self-report using the State Energy and Fatigue Scale. There are 3 items, scored using a number line from 0 to 100, that are summed to generate a score, where higher scores indicate greater mental fatigue.
Physical Energy | Before and immediately after stair walking
  Measured by self-report using the State Energy and Fatigue Scale. There are 3 items, scored using a number line from 0 to 100, that are summed to generate a score, where higher scores indicate greater physical energy.
Physical Fatigue | Before and immediately after stair walking
  Measured by self-report using the State Energy and Fatigue Scale. There are 3 items, scored using a number line from 0 to 100, that are summed to generate a score, where higher scores indicate greater physical fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Gay, PhD, Principal Investigator — University of Georgia
Locations (1):
- Ramsey Center, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, data may be shared for primary and secondary outcomes.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Upon publication of the primary and secondary outcomes
Access Criteria: Data access requests will be reviewed by the study team. Requestors will be required to sign a Data Access Agreement.